CLINICAL TRIAL: NCT04548934
Title: Effect of Wearing Personal Protective Equipment (PPE) on CPR Quality in Times of the COVID-19-pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPR PPE
Record Dates: First submitted 2020-09-02; First posted 2020-09-16 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-09

CONDITIONS: Cardiopulmonary Resuscitation; Personal Protective Equipment
MeSH Terms: interventions — Personal Protective Equipment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No PPE (Active Comparator): Cardiopulmonary resuscitation without wearing personal protective equipment (PPE)
  Interventions: Device: No Personal protective equipment (PPE)
- PPE (Experimental): Cardiopulmonary resuscitation while wearing personal protective equipment (PPE)
  Interventions: Device: Personal protective equipment (PPE)

INTERVENTIONS:
Device: Personal protective equipment (PPE) — Wearing of PPE (FFP3 mask, gloves, eye protection, long-sleeved gown)
  Arms: PPE
Device: No Personal protective equipment (PPE) — Standard CPR without wearing PPE
  Arms: No PPE

SUMMARY:
Background The significant risk of transmission of SARS-CoV-2 to healthcare staff mandated changes to Basic and Advanced Life Support (BLS and ALS) guidelines. As advised by the European Resuscitation Council (ERC), healthcare staff should put on airborne-precaution personal protective equipment (PPE) before starting chest compressions and/or airway interventions, as a minimum an FFP3 mask (FFP2 or N95 if FFP3 not available), eye and face protection and long-sleeved gown. However, wearing FFP3 masks has been shown to highly impair cardiopulmonary exercise capacity and the effect of wearing PPE on the quality of cardiopulmonary resuscitation is not known. The aim of this project is therefore to to investigate whether wearing PPE has an effect on the quality of chest compressions.

Methods The study forsees a simulated CPR scenario on manikins. Study participants are lay rescuers and members of the rescue organization Croce Bianca. Each participant will perform 5 sequences consisting of 2 min of chest compressions altered by 2 min of no chest compressions (break), as recommended by the current ERC guidelines. The participants will perform the described CPR sequence two times in a cross-over design with randomized order, once while wearing PPE and once without wearing PPE. Between the two CPR sequences (i.e. with and without PPE) a break of 60 min for recovery will be given. During both CPR sequences, the quality of chest compressions will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Member of the rescue organization "Croce Bianca"
* Aged 18-60
* Certified in basic life support (BLS)
* No current COVID-19 symptoms, not being tested positive for COVID-19, no COVID-19 symptoms in the 4 weeks before the tests, no quarantine or unprotected contacts with COVID positive patients in the last 4 weeks, body temperature ≤ 37.5°on test days.
* Obtained informed consent.

Exclusion Criteria:

* Age <16 or >60 years,
* No informed consent
* Current COVID-19 symptoms, being tested positive for COVID 19 or symptoms in the 4 weeks before the tests, quarantine or unprotected contacts with COVID-19 positive patients in the last 4 weeks, body temperature ≥ 37.5°on test days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Depth of chest compression | 20 minutes of CPR
  Difference in chest compression depth during a simulated cardio-pulmonary resuscitation (CPR) on manikins when performed with and without wearing personal protective equipment (PPE).

SECONDARY OUTCOMES:
Chest compression rate | 20 minutes of CPR
  Difference in chest compression rate during a simulated cardio-pulmonary resuscitation (CPR) on manikins when performed with and without wearing personal protective equipment (PPE).
Relaxation | 20 minutes of CPR
  Difference in the percentage of compressions with incomplete release during a simulated cardio-pulmonary resuscitation (CPR) on manikins when performed with and without wearing personal protective equipment (PPE).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rauch, MD, PhD, Principal Investigator — Eurac research, Institute of mountain emergency medicine
Locations (1):
- Headquarter of "Croce Bianca" EMS organization, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: No